CLINICAL TRIAL: NCT00790075
Title: Liquid Risperidone in the Treatment of Acute Agitation in Psychiatrically Hospitalized Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Gabrielle A. Carlson, MD, StonyBrook University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20034920
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Agitation
Keywords: agitation; Episodes of agitation regardless of diagnosis
MeSH Terms: conditions — Psychomotor Agitation | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: risperidone — liquid risperidone was administered on a mg/kg basis to a child needing seclusion. 0.015mg/kg was the start dose. Dose was increased to 0.02mg/kg if duration of episode was >30 minutes.

SUMMARY:
The goal of this study is to demonstrate safety and efficacy of liquid risperidone in psychiatrically hospitalized children, ages 4-12, who would be put in seclusion or restraint, or given an intramuscular injection of diphenhydramine because of their out-of-control behavior if not medicated with risperidone. The first part of the study will: 1) develop appropriate oral doses of medication to reduce out of control or agitated behavior effectively with the fewest side effects, and 2) develop a rating system to measure the children's behavior i.e. level of improvement, sedation, and untoward effects.

DETAILED DESCRIPTION:
A. Develop an appropriate dose structure for risperidone. Children needing oral medication will be initially offered a safe minimal dose (0.015 mg/kg) dose of risperidone (between 0.3 and 0.6mg for children weighing between 20-40kg). If there is no response, or an inadequate response (anything less than "much improved" on the Clinical Global Improvement Scale) after 30 minutes, the next dose (0.02 mg/kg) will be used if there is another occasion to use a medication intervention the following day. Similarly, a medium dose (0.025 mg/kg) dose will be used if the lower dose is inadequate. The highest dose is 0.3mg/kg. For a big child (we have had children who weigh as much as 55kg this would work out to a maximum dose of 1.6 mg/dose, well within the dose range administered on a one time, daily basis to children (2 mg is the usual maximum, though a daily dose of 3-4 mg is not uncommon). If the child is already receiving risperidone, total daily dose will not exceed 0.07mg/kg/day (the maximum dose used in the RUPP trial). Weight dose chart follows on the next page. Intervention following the 30 minutes will depend on clinical judgement. It may include a different medication, open seclusion, or room restriction.

B. Develop a rating instrument for the stages of agitation needing to be rated. It has been difficult to operationalize when to intervene, and how to rate improvement. There are absolutely no guidelines on this. We have developed a list of behaviors that a nurse rater will use to observe the child at 5, 15, 30, 45, 60, 90 and 120 minutes after any intervention for an episode of agitation. We will, of course, be specifically interested in these measures for children receiving risperidone. (It maybe necessary to videotape some children to develop reliability on the measure.) The advantage of using such an instrument will be that the children will be very closely observed for both positive and negative effects. However, in short term treatment trials, sedation and fatigue were the most common "adverse event", followed by increased appetite. Neurologic side effects (tremor, dyskinesia, rigidity, akathesia and difficulty swallowing) have been reported in chronic use of this medication in adults. In children, in the placebo controlled study, only tremor was marginally more common in the risperidone group.

We anticipate having about 20 children and about 60 episodes of severe agitation over a 9 month period during which we will be able to find a reasonable dose of risperidone, determine its onset and duration of action, and its efficacy in shortening episodes of severe agitation.

INCLUSION AND EXCLUSION CRITERIA All psychiatrically hospitalized children on 12North who are unable to take a "time out" because they are agitated and out of control are eligible for this study. These are children who ordinarily would be treated either with seclusion/restraint or an intra-muscular shot of diphenhydramine (Benadryl). Excluded children would be those who have had allergic or "bad" reactions to risperidone in the past, and those in whom adequate doses have not produced improvement in behavior. Since liquid risperidone is frequently used as an intervention on the unit anyway, being part of this study is, in fact providing closer supervision than is usually undertaken. Close supervision is not required for safety and we are doing it as part of this project to more precisely document onset and offset of medication effect as well as to establish a pattern of symptom remission.

RISKS AND DISCOMFORTS The side effects that most frequently occurred in children treated every day for several months with this medication include increased appetite, weight gain, feeling tired and drowsy, tremor and dyskinesia. Long term use is most associated with weight gain. There is a very small risk of extrapyramidal symptoms (akathesia, dystonia). This is usually seen with doses higher than are used in this study, but may occur. Prolactin elevation and galactorrhea rarely occur, but also are most associated with long term use.

BENEFITS Development of a safe and effective treatment for severe agitation in children. Development of a rating scale that can be used in other intervention studies. We reiterate that this intervention is used in children without very much information so the close supervision following treatment may also be a benefit.

ELIGIBILITY:
Inclusion Criteria:

* consented, psychiatrically hospitalized child between the ages of 4-12 whose agitated behavior would otherwise require seclusion

Exclusion Criteria:

* prior side effects taking risperidone

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2003-01; Primary Completion 2004-06 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
reduced time to end of agitation episode compared to unmedicated agitation episode | Duration of "time out" or time in seclusion

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle A Carlson, MD, Principal Investigator — StonyBrook University School of Medicine
Locations (1):
- StonyBrook University Hospital (StonyBrook University School of Medicine), Stony Brook, New York, United States